CLINICAL TRIAL: NCT03429504
Title: Impact of Body Mass Index on Outcomes of Breast Cancer Management (Retrospective Study)
Brief Title: Impact of Body Mass Index on Outcomes of Breast Cancer Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moheb Ibrahim Melek, Principal Investigator, Assiut University
Other Study IDs: BMIBC
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Obesity and Breast Cancer
Keywords: Obesity; Breast cancer; Body mass index
MeSH Terms: conditions — Obesity; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese breast cancer patients: Response to treatment and progression free survival in obese breast cancer patients
- non obese breast cancer patients: Response to treatment and progression free survival in non obese breast cancer patients

SUMMARY:
Obesity has been linked to an increased risk of developing a number of malignancies, including postmenopausal breast cancer. One of the established risk factors for breast cancer development in post-menopausal women is obesity which has further been linked to breast cancer recurrence and poorer survival in pre- and post-menopausal breast cancer.

DETAILED DESCRIPTION:
The biological mechanisms underlying the association between obesity and breast cancer could involve interacting mediators of hormones, adipocytokines, and inflammatory cytokines which link to cell survival or apoptosis, migration and proliferation. Higher level of oestradiol produced in postmenopausal women through aromatization of androgens in the adipose tissues and higher level of insulin, a condition common in obese women, are linked to poorer prognosis in breast cancer. A possible interaction between leptin, insulin and obesity-related markers of inflammation have also been linked to breast cancer outcomes. Non-biological mechanisms could include chemotherapy under-dosing in obese women, suboptimal treatment, and obesity-related complications.

The impact of body mass index on treatment outcome in patients receiving endocrine therapy, there have been consistent results indicating that the efficacy of aromatase inhibitors vary with body mass index; however, the efficacy of tamoxifen is not body mass index-dependent. In the Arimidex, Tamoxifen, Alone or in Combination trial, which compared the efficacy of anastrozole against tamoxifen as an adjuvant treatment for hormone receptor-positive post-menopausal breast cancer patients, anastrozole, a non-steroidal aromatase inhibitor, was significantly less effective in post-menopausal breast cancer patients with a high body mass index, whereas an equal efficacy of tamoxifen was shown across all body mass index levels.

Observational study. Retrospective analysis of data that will be collected from breast cancer patients medical records as body mass index and their response to treatment, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Medical records of female Patients with breast cancer at clinical oncology and nuclear medicine department, Assiut University Hospital between (1st Jan 2012 and 31st Dec 2016), their recorded body mass index and their follow up will be included in the study.

Exclusion Criteria:

* Patients' medical records that had no documented weight and height.
* Patients' medical records that had no documented follow up.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer that was admitted at clinical oncology and nuclear medicine department, Assiut University Hospital, Egypt
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-12 (Estimated); Primary Completion 2019-02-12 (Estimated); Study Completion 2019-08-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of obese breast cancer patients with response to treatment compared to non obese breast cancer patients. | The cases will be obtained from the medical records of breast cancer patients admitted to the Clinical Oncology and Nuclear Medicine Department, Assiut University hospital from 1st of January, 2012 - 31st December, 2016

CONTACTS AND LOCATIONS:
Overall Officials: Aiat M Mohamed, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deglise C, Bouchardy C, Burri M, Usel M, Neyroud-Caspar I, Vlastos G, Chappuis PO, Ceschi M, Ess S, Castiglione M, Rapiti E, Verkooijen HM. Impact of obesity on diagnosis and treatment of breast cancer. Breast Cancer Res Treat. 2010 Feb;120(1):185-93. doi: 10.1007/s10549-009-0459-1. Epub 2009 Jul 14. PMID 19597985
- [Background] Yung RL, Ligibel JA. Obesity and breast cancer: risk, outcomes, and future considerations. Clin Adv Hematol Oncol. 2016 Oct;14(10):790-797. PMID 27930630
- [Background] Protani M, Coory M, Martin JH. Effect of obesity on survival of women with breast cancer: systematic review and meta-analysis. Breast Cancer Res Treat. 2010 Oct;123(3):627-35. doi: 10.1007/s10549-010-0990-0. Epub 2010 Jun 23. PMID 20571870
- [Background] Ligibel J. Obesity and breast cancer. Oncology (Williston Park). 2011 Oct;25(11):994-1000. PMID 22106549
- [Background] Niraula S, Ocana A, Ennis M, Goodwin PJ. Body size and breast cancer prognosis in relation to hormone receptor and menopausal status: a meta-analysis. Breast Cancer Res Treat. 2012 Jul;134(2):769-81. doi: 10.1007/s10549-012-2073-x. Epub 2012 May 5. PMID 22562122
- [Background] Sestak I, Distler W, Forbes JF, Dowsett M, Howell A, Cuzick J. Effect of body mass index on recurrences in tamoxifen and anastrozole treated women: an exploratory analysis from the ATAC trial. J Clin Oncol. 2010 Jul 20;28(21):3411-5. doi: 10.1200/JCO.2009.27.2021. Epub 2010 Jun 14. PMID 20547990